CLINICAL TRIAL: NCT01892787
Title: Randomised Controlled Single and Chronic Dosing Crossover Comparison of Extra Fine Particle Formoterol and Coarse Particle Salmeterol in Asthmatic Patients With Persistent Small Airways Dysfunction
Brief Title: Effects of Particle Size in Small Airways Dysfunction
Acronym: MAN03
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor of Allergy and Pulmonolgy, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013RC01; 2013-001103-36 (EudraCT Number); 13/ES/0050 (Other: East of Scotland Research Ethics Service REC2)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: Asthma; Small airways; Extra fine particle long-acting beta agonists
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formoterol (Atimos Modulite) (Experimental): Atimos Modulite 1 puff (12 micrograms) twice a day
  Interventions: Drug: Formoterol
- Salmeterol (Serevent Accuhaler) (Active Comparator): Serevent Accuhaler 1 puff (50 micrograms) of twice a day
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Formoterol — Participants receive Atimos for 1 to 2 weeks.Partcipants then enter a washout period and after the washout period receive the alternative treatment arm.
  Other Names: Atimos Modulite
  Arms: Formoterol (Atimos Modulite)
Drug: Salmeterol — Participants receive Serevent for 1 to 2 weeks. Participants then enter a washout period and after the washout period receive the alternative treatment arm.
  Other Names: Serevent Accuhaler
  Arms: Salmeterol (Serevent Accuhaler)

SUMMARY:
The airways in the lungs get smaller the further into the lungs they go. Most simple measurements of lung function only reflect the larger 'central' airways and do not provide information on the smaller 'peripheral' airways. Newer measurements have been developed that can now give us accurate information on how the smaller airways are working. Indeed the small airways seem to play a significant role in asthma in terms of inflammation and airway narrowing. Recently, new types of inhaler formulations have been developed that have a much smaller particle size than other standard formulations. These formulations have been shown to go further into the lungs, thus getting into the smaller airways. In this study we aim to compare the two extremes of available long acting beta agonists in terms of particle size i.e. extra fine formoterol (Atimos) versus coarse particle salmeterol (Serevent)in asthmatics with abnormal small airway function using a breathing test called impulse oscillometry. By using this test we will be able to find out whether using an extrafine particle inhaler improves small airway function.

DETAILED DESCRIPTION:
The small airways are gaining greater recognition for their role in the pathophysiology of persistent asthma and as a relevant target for asthma treatment(1). Pathological abnormalities in the small airways have been demonstrated regardless of asthma severity and seem to persist even in patients with stable asthma(2, 3).

Historically, the small airways have been difficult to assess. Spirometry generally reflects large airways function although the mean forced expiratory flow (FEF) between 25% and 75% of FVC (FEF25-75) has been used to assess small airway obstruction.(4) More recently, impulse oscillometry (IOS) has been used to assess the role of small airways in asthma(5). IOS is an effort-independent test, using oscillation of differing sound waves to derive a variety of output measurements determining both the degree of total and peripheral airway resistance. Resistance at 5 Hz reflects total airway resistance and central airway resistance is approximated using resistance at 20 Hz (R20). The peripheral or small airway component can thus be evaluated by calculating the difference between these two measurements i.e. R5 - R20.

We have identified from our database of primary care referrals, a cohort of patients who appear to have evidence of an unmet physiological need in terms of persistent small airways dysfunction, on the basis of impairment of R5 and R5-R20 despite taking step 2/3/4 asthma treatment(6). Approximately 32% of patients across steps 2/3/4 had severely abnormal values for both R5-R20 (>0.05 kPa/L.s) and R5 (> 150%). Such small airway dysfunction at step 3/4 occurred despite patients being prescribed ICS with LABA, although there were no patients being prescribed extra fine ICS/LABA or extra fine LABA (i.e. Fostair or Atimos). In terms of the ICS moiety, observational data has shown that patients taking extra fine HFA-beclometasone solution (Qvar) have equal or better control than those taking Fluticasone suspension, while receiving a lower maintenance dose of ICS(7). In another study, patients switched from beclometasone suspension to solution at half the dose had an improvement in asthma quality of life. In neither of these studies was there any information available regarding small airway dysfunction in order to explain the potential improvements with HFA-beclometasone(8).

There is a paucity of information on the potential benefits of extra fine formoterol on the small airways. In a single dosing study comparing extra fine HFA versus coarse particle dry powder formulations of formoterol, there was a 30% difference (absolute difference of 2.9 kPa/L.s.min)in R5 AUC0-60min and 63% difference (absolute difference of 2.4 kPa/L.s.min) in R5-R20 AUC0-60min, although this was not the primary end point(9).

1.2 RATIONALE Thus, the primary objective for the present study is to compare the two extremes of available long acting beta-agonist formulations - i.e. extra fine HFA formoterol ( Atimos ) versus coarse particle DPI salmeterol (i.e. Serevent Accuhaler). If there turns out to be a significant improvement in small airways function conferred by extra fine formoterol, then this would in turn support the rationale for performing a further chronic study to assess the clinical impact of treating persistent small airways dysfunction at step 3/4 by switching patients to Fostair HFA and comparing to Seretide DPI, in terms of improving asthma control in patients with the small airway phenotype who are already taking conventional ICS/LABA formulations. We will use impulse oscillometry to assess the small airways response using the difference between resistance measured at 5Hz and 20Hz (R5-R20) as the primary outcome. In this regard we have previously reported in asthmatic patients receiving propranolol that there was a 104.1 % (95%CI 22.6-185.6%) worsening of R5-R20 in terms of the bronchoconstrictor response to propranolol, and following subsequent histamine challenge, there was a 115.6 % (95%CI 55.6-175.7% ) improvement in R5-R20 in terms of the bronchodilator response to nebulised salbutamol.(10)

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers aged at least 16 years with a diagnosis of asthma
* Persistent severe small airways dysfunction on impulse oscillometry with R5 > 150% and R5-R20 > 0.05 kPa/L.s despite taking ICS or inhaled corticosteroids / long-acting beta-agonists
* FEV1 > 60 %
* Ability to give informed consent
* Agreement for their GP to be made aware of study participation and to receive feedback as relevant to the participant's well being

Exclusion Criteria:

* Participants already receiving extra-fine particle long-acting beta agonists
* Other respiratory diseases such as chronic obstructive pulmonary disease, bronchiectasis or alergic allergic bronchopulmonary aspergillosis
* An asthma exacerbation or respiratory tract infection requiring systemic steroids and/or antibiotics within 3 months of the study commencement
* Smoking within one year or 10 pack year history
* Any clinically significant medical condition that may endanger the health or safety of the participant
* Participation in another trial within 30 days before the commencement of the study
* Pregnancy or lactation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in R5-R20 as change from baseline after first and last dose | At baseline & after 1-2 weeks
  R5 - Resistance at 5Hz, R20 - Resistance at 20Hz

SECONDARY OUTCOMES:
Change in remaining impulse oscillometry variables (R5,R20,X5,AX,RF) after first and last dose | Baseline and after 1-2 weeks
  R5 - Resistance at 5Hz, R20 - Resistance at 20Hz, X5 - Reactance at 5Hz, RF - Frequency of resonance, AX - Area under reactance curve
Area under the curve from 0 to 60 min | Baseline and 1-2 weeks
Spirometry | Baseline & 1-2 weeks
  Forced expiratory volume in 1 second (FEV1); forced vital capacity (FVC); forced expriatory flow between 25-75% of vital capacity.
Domiciliary peak expiratory flow | 1-2 weeks
Asthma Control Questionnaire | 1-2 weeks
Exhaled nitirc oxide | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lipworth, MD, Principal Investigator — University of Dundee; Arvind Deva Manoharan, MBChB, Principal Investigator — University of Dundee
Locations (1):
- Brian Lipworth, Dundee, United Kingdom

REFERENCES:
- [Result] Manoharan A, von Wilamowitz-Moellendorff A, Morrison A, Lipworth BJ. Effects of formoterol or salmeterol on impulse oscillometry in patients with persistent asthma. J Allergy Clin Immunol. 2016 Mar;137(3):727-33.e1. doi: 10.1016/j.jaci.2015.06.012. Epub 2015 Jul 26. PMID 26220533